CLINICAL TRIAL: NCT00973206
Title: Factors Influencing Cardiovascular Prognosis in Hypertensive Patients (Pythia Study)
Brief Title: Factors Influencing Cardiovascular Prognosis
Acronym: Pythia-GR
Status: Not yet recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vasilios Kotsis, Prof. Med, Aristotle University Of Thessaloniki
Other Study IDs: AUTH20090609
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Cardiovascular Mortality
Keywords: cardiovascular morbidity; mortality community study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify risks for cardiovascular events in a follow up period of 10 years.

DETAILED DESCRIPTION:
Inclusion criteria

* Age > 50 years volunteers (2 towns of 15000 residents one in the north and one in the south of Greece)
* End points
* 5-10 years cardiovascular morbidity and mortality

Measurements at baseline

* Anthropometrics

  * Age (M>55 years; W>65 years)
  * Weight-height- BMI
  * Abdominal obesity (Waist circumference>102 cm(M), >88cm (W) Family history
  * Family history of premature CV disease (M at age<55 years; W at age<65 years)

History

* Smoking
* Diabetes Mellitus,
* Established Heart disease: myocardial infarction; angina; coronary revascularization; heart failure
* Established renal disease [diabetic nephropathy; renal impairment (serum creatinine M>133, W>124 mmol/l); proteinuria (> 300 mg/24 h)]
* Cerebrovascular disease: ischaemic stroke; cerebral haemorrhage; transient ischaemic attack
* Peripheral artery disease
* Advanced retinopathy: haemorrhages or exudates, papilloedema
* Treatment

Measurements

* Measurements Blood pressure

  * Clinic BP
  * 24h ABPM
  * Home BP

Heart

* Electrocardiographic LVH
* Echocardiographic LVH

Vessels

* Carotid wall thickening or plaque
* Carotid-femoral pulse wave velocity
* Ankle/brachial BP index

Lipids or other risk factors

* Total cholesterol, Tg, HDL, LDL
* Plasma creatinine, estimated glomerular filtration rate
* Fasting plasma glucose or postload plasma glucose
* Microalbuminuria and albumin-creatinine ratio
* Glucose tolerance test

  * Follow up each 3 year with all the above measurements

ELIGIBILITY:
Inclusion Criteria:

* All age >50 volunteers

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers,community sample, residents of a certain town
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 10 years

SECONDARY OUTCOMES:
Hospitalization for CV events | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Kotsis, Prof, Study Chair — AUTH